CLINICAL TRIAL: NCT03499561
Title: a Symptomatic Bacteriuria in Pregnant Females
Brief Title: a Smptomatic Bacteriuria in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Assistant Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: A symptomatic bacteriuria
Record Dates: First submitted 2018-04-06; First posted 2018-04-17 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Bacteriuria in Pregnancy
MeSH Terms: interventions — Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- pregnant women in first Trimester: A urine sample will be taken from pregnant women before 14 weeks of pregnancy
  Interventions: Diagnostic Test: urine analysis
- pregnant women in second Trimester: A urine sample will be taken from pregnant women from 14 weeks +1 day till 28 weeks
  Interventions: Diagnostic Test: urine analysis
- pregnant women in third Trimester: A urine sample will be taken from pregnant women from 28 weeks +1 day till 40 weeks
  Interventions: Diagnostic Test: urine analysis

INTERVENTIONS:
Diagnostic Test: urine analysis — Intervention is (urine analysis ): of a mid stream urine sample will be taken

SUMMARY:
Asymptomatic bacteriuria (ASB) is defined as the presence of at least 105 colony-forming units (CFU)/ml of 1 or 2 bacterial species in clean-voided midstream urine sample from an individual without symptoms of UTI

DETAILED DESCRIPTION:
ASB is common in women and increases in prevalence with age and/or sexual activity, due to short urethra, pregnancy, easy contamination of urinary tract with fecal flora

The pregnant women are two times more commonly affected than age matched non pregnant females. This is due to urinary stasis due to progesterone effect in pregnancy in addition to different morphological and physiological changes occurring during pregnancy The prevalence of ASB is about 3 times higher in diabetic women (ranging from 15% to 30%) than in non-diabetic women (less than 10%)

ELIGIBILITY:
Inclusion Criteria:

* 1. Pregnant females 2. Non-symptomatic females.

Exclusion Criteria:

* 1. Patients taking antibiotics in the last two weeks. 2. Symptomatic UTI. 3. Suspected urinary tract abnormalities. 4. Urinary catheterization. 5. Renal dialysis.

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — pregnant females with no symptoms
Study Population: Pregnant non-symptomatic females.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
The number of participants who will discovered to have bacteriuria | within 4 weeks
  Incidence of asymptomatic bacteriuria among pregnant females.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
The research will be published after finishing results